CLINICAL TRIAL: NCT02446275
Title: DO SOFT TISSUE TECHNIQUES HAVE A POSITIVE EFFECT ON DISABILITY AND QUALITY OF LIFE IN MIGRAINE SUFFERERS?: A Randomized Controlled Trial
Brief Title: Efficacy of Manual Therapy in Migraine
Acronym: MTHDIQMi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PT, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID005
Record Dates: First submitted 2015-03-20; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: MIGRAINE
Keywords: efficacy, manual therapy, migraine, quality of life
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sternocleidomastoid MTRP and stretching (Experimental): The sternocleidomastoid was treated with ischemic compression.
  Interventions: Other: Trapezius MTRP and stretching
- Trapezius MTRP and stretching (Experimental): The central MTRP of the trapezius was treated as described above for the sternocleidomastoid.
  Interventions: Other: Sternocleidomastoid MTRP and stretching

INTERVENTIONS:
Other: Sternocleidomastoid MTRP and stretching — The sternocleidomastoid was treated with ischemic compression. The patient's head was passively moved into contralateral rotation and the patient was asked to relax completely. Sustained pressure was then applied to the sternocleidomastoid muscle until the pain threshold was reached. During the application of pressure, pain decreases so the pressure was gradually increased over a duration of 1 minute. The pressure was then reduced progressively.
  Arms: Trapezius MTRP and stretching
Other: Trapezius MTRP and stretching — The central MTRP of the trapezius was treated as described above for the sternocleidomastoid. Subsequently stretching was performed, whereby the therapist supported the patient's head and performed passive contralateral inclination and ipsilateral rotation of the head. The therapist placed one hand over the patients shoulder while the other hand performed the stretching and simultaneously controlled the position of the head to achieve suitable stretching
  Arms: Sternocleidomastoid MTRP and stretching

SUMMARY:
Objective: The aim of this study was to determine the efficacy of suboccipital inhibitory manual therapy treatment in migraine compared to treatment based on Myofascial Trigger Points (MTrPs) and their stretching, often being hypersensitive in patients with migraine.

Material and methods: 27 patients in two groups participated in the study: a) the control group received combined techniques based on MTrPs and bilateral stretching in the trapezius and sternocleidomastoid muscle (SCM); b) the experimental group was applied the same techniques as those applied in the control group plus suboccipital inhibition. The treatment lasted for 8 weeks and the impact, disability and quality of life were assessed in both groups.

DETAILED DESCRIPTION:
Introduction Migraine is a highly prevalent disorder entailing substantial costs. Manual therapy offers an attractive option as an alternative to medical treatment or used in combination therewith. Treatment focused on the soft tissues of the suboccitpital region has been studied in other types of headaches but not in migraine.

Objective: The aim of this study was to determine the efficacy of suboccipital inhibitory manual therapy treatment in migraine compared to treatment based on Myofascial Trigger Points (MTrPs) and their stretching, often being hypersensitive in patients with migraine.

Material and methods: 27 patients in two groups participated in the study: a) the control group received combined techniques based on MTrPs and bilateral stretching in the trapezius and sternocleidomastoid muscle (SCM); b) the experimental group was applied the same techniques as those applied in the control group plus suboccipital inhibition. The treatment lasted for 8 weeks and the impact, disability and quality of life were assessed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed according to the criteria established by the IHS

Exclusion Criteria:

* Patients were excluded if they presented with other headache types, if their headache was triggered by neck movement, or if they presented with dizziness, hypertension, emotional stress, psychological disorders, cardiovascular disease or pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  The Visual Analogue Scale (VAS)25 was used to rate the patients average pain intensity using a 0-10 scale (0=no pain, 10=the most severe pain).

SECONDARY OUTCOMES:
The impact of headache (HIT-6) | 4 weeks
  The Headache Impact Test (HIT-6) (Yang et al., 2011) provides an overall measure of the adverse impact of headaches. This questionnaire consists of 6 items measuring the impact of pain on social functioning, role functioning, vitality, cognitive functioning and psychological distress, and provides a measure of the severity.
Disability (MIDAS) | 4 weeks
  . Disability caused by migraine was assessed by the MIDAS questionnaire (Adenis Silva et al., 2008) based on 5 questions and the score obtained from the sum of the days lost due to headaches registered in the questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma v. Espí López, Valencia, Valencia, Spain

REFERENCES:
- [Background] Fernandez-de-las-Penas C, Dommerholt J. Myofascial trigger points: peripheral or central phenomenon? Curr Rheumatol Rep. 2014 Jan;16(1):395. doi: 10.1007/s11926-013-0395-2. PMID 24264721
- [Background] Becker C, Brobert GP, Almqvist PM, Johansson S, Jick SS, Meier CR. Migraine incidence, comorbidity and health resource utilization in the UK. Cephalalgia. 2008 Jan;28(1):57-64. doi: 10.1111/j.1468-2982.2007.01469.x. Epub 2007 Nov 6. PMID 17986274
- [Background] Calandre EP, Hidalgo J, Garcia-Leiva JM, Rico-Villademoros F. Trigger point evaluation in migraine patients: an indication of peripheral sensitization linked to migraine predisposition? Eur J Neurol. 2006 Mar;13(3):244-9. doi: 10.1111/j.1468-1331.2006.01181.x. PMID 16618340